CLINICAL TRIAL: NCT04377854
Title: The Prognostic Value of proBNP in Patients Supported With Durable Mechanical Circulatory Assist Devices - a 25 Year Follow up Study.
Brief Title: Prognostic Value of BNP in MCS - a 25 Year Follow up Study
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Finn Gustafsson, Professor, Rigshospitalet, Denmark
Other Study IDs: H-19055497
Record Dates: First submitted 2020-05-03; First posted 2020-05-06 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure; Left Ventricular Assist Device; Prognosis; Durable Mechanical Support Device
MeSH Terms: conditions — Heart Failure | interventions — Observation; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MCS recipients: All recipients of durable MCS will be followed up on a yearly basis with collection of blood sample and clinical data for 25 years.
  Interventions: Other: 2) Observation and collection and of blood sample
- Recipient of cardiac transplant: All recipients of cardiac transplantation(s) will be followed up on a yearly basis with collection of clinical data for 25 years.
  Interventions: Other: Observation. No intervention per se.
- Watchful waiting at Rigshospitalet: Patients referred for evaluation for treatment with advanced treatment (LVAD/HTX) but -for whatever reason- these pts will be on watchful waiting at the Rigshospitalet.
  Interventions: Other: Observation. No intervention per se.

INTERVENTIONS:
Other: Observation. No intervention per se. — Observation. No intervention (no collection of blood).
  Other Names: 1) Observation - No intervention
  Groups: Recipient of cardiac transplant; Watchful waiting at Rigshospitalet
Other: 2) Observation and collection and of blood sample — All patients evaluated for adv HF (HTX/LVAD) will be offered to contribute to this database; Blood samples will be collected from all at baseline. Patients receiving LVAD will contribute on a yearly basis (or until withdrawal of consent). For other patients no further blood will be collected unless they receive an LVAD at a later point.
  Other Names: Blood sample
  Groups: MCS recipients

SUMMARY:
A biobank has been created to investigate the prognostic value of biomarkers (mainly BNP) in patients implanted with durable mechanical assist devices comparing patients with advanced HF supported by MCS with those who are transplanted and those who remain on optimal medical therapy.

Patients will be followed up for 25 years after inclusion.

DETAILED DESCRIPTION:
All patients referred for advanced HF treatment at the Dept of Cardiology at Rigshospitalet.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for evaluation for advanced HF treatment at the Rigshospital in Denmark
* Age>18 years

Exclusion Criteria:

* No consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients referred for evaluation for advanced HF treatment at the Rigshospitalet in Denmark. All patients with Advanced HF (regardless of type of adv HF treatment) at the contributing center will (hopefully) be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-18 (Actual); Primary Completion 2045-08-01 (Estimated); Study Completion 2045-08-01 (Estimated)

PRIMARY OUTCOMES:
Alive | 25 years from inclusion
Dead | 25 years from inclusion
  Dead after inclusion in study

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, DK, Denmark

IPD SHARING:
Plan to Share IPD: No